CLINICAL TRIAL: NCT05905302
Title: The Impact of Exercise on Subthalamic Nucleus Neural Activity in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jay Alberts (Other)
Responsible Party: Sponsor-Investigator, Jay Alberts, Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R21NS129147-01 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Fifteen Parkinson's disease patients who have undergone DBS surgery and utilize the Percept system will complete a FE and VE exercise session on a stationary cycle while OFF antiparkinsonian medication. Bilateral neural activity of the STN will be continuously recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Two modes of high intensity exercise
  Interventions: Other: Forced and Voluntary Exercise

INTERVENTIONS:
Other: Forced and Voluntary Exercise — Participants will complete a forced exercise (FE) and voluntary exercise (VE) session. Forced exercise is a mode of high intensity exercise in which voluntary exercise rate is augmented, but not replaced. Voluntary exercise is standard stationary cycling. FE and VE exercise sessions will be Off antiparkinsonian medication. The order in which exercise session is conducted first will be randomized. Bilateral neural activity of the STN will be continuously recorded for 130 minutes (pre, during FE or VE and post-exercise).

SUMMARY:
Fifteen PwPD who have undergone DBS surgery and utilize the Percept system will complete a FE and VE exercise session on a stationary cycle while Off antiparkinsonian medication. Bilateral neural activity of the STN will be continuously recorded for 130 minutes (pre-, during FE or VE and post-exercise). The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III Motor Exam and upper extremity force-tracking task will be used to determine motor response to exercise.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurological disease, most prevalent in older adults, estimated to affect over 12 million people world-wide by 2040. While antiparkinsonian medication and deep brain simulation (DBS) are effective in managing disease symptoms, disease modification has remained elusive. Exercise has been proposed as the Universal Prescription for PD capable of slowing disease progression; stationary cycling in particular has been suggested as an ideal exercise modality for people with PD (PwPD).Our seminal tandem cycling study was the first to utilize forced exercise (FE) in human PD patients and demonstrate a 30% improvement in clinical ratings compared to voluntary exercise (VE). Briefly, FE is a mode of high intensity exercise originating in animal models of PD in which voluntary exercise rate is augmented, but not replaced. Thus, PwPD were assisted in pedaling at a higher rate (cadence) on the tandem cycle compared to those on a standard stationary cycle performing voluntary exercise (VE). This work resulted in a paradigm shift in terms of recommending high intensity exercise for PwPD. Currently, we are involved in two multi-site clinical trials aimed at identifying the potential of high intensity exercise to slow PD (2R01NS073717 & 1U01NS113851). Despite the potential of exercise to alter disease progression, its mechanism of action and effects on basal ganglia function are not understood. The loss of dopamine producing neurons associated with PD results in hypersynchrony of basal ganglia motor circuits that underlies PD symptoms. Recent animal studies using FE evaluated neural activity, local field potentials (LFPs), from the primary motor cortex (M1) to estimate the impact of exercise on basal ganglia function. Following FE, neural hypersynchrony in the beta (13-35Hz) frequency band was reduced in M1, which was proposed to underlie improved motor function. M1 activity is impacted by the activity in the subthalamic nucleus (STN), a structure in the basal ganglia, via the direct and indirect pathways. The impact of high intensity exercise, VE or FE, on STN hypersynchrony in humans is unknown. Recording of STN neural activity, until recently, was only possible during DBS surgery or in patients whose electrode was temporarily externalized immediately post-surgery. Neither approach is feasible or safe to systematically evaluate the effects of exercise on basal ganglia function. Recently, the Medtronic Percept DBS platform received FDA approval. The Percept platform records and streams neural activity from the DBS electrode within the STN. This project, for the first time, will record neural activity from the STN during two modes of high intensity exercise, FE and VE, in PwPD to identify the potential mechanism underlying the beneficial effects of exercise on PD. Our underlying hypothesis is that high intensity exercise reduces STN hypersynchrony which facilitates cortico-basal ganglia-thalamocortical circuit functionality thereby improving motor function following exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with a diagnosis of PD by a movement disorders neurologist
2. Previous placement, at least six months, of bilateral Medtronic Precept DBS as standard of care treatment for their PD.
3. Stable and clinically optimized DBS parameters for three months prior to enrollment.
4. Demonstrate the ability to safely mount and dismount a recumbent exercise cycle with an upright back.
5. Willingness to withhold antiparkinsonian medication and DBS stimulation.
6. Exercise clearance using the American College of Sports Medicine (ACSM) Pre-participation Health Screen: a. If the ACSM screen recommends medical clearance, the subject must obtain medical clearance by their health care provider prior to participation; b. Those who choose not to obtain physician clearance will not be eligible for participation.

Exclusion Criteria:

1. Diagnosis of dementia or any neurocognitive impairment that compromises the ability to provide informed consent.
2. A musculoskeletal issue that limits one's ability to cycle
3. Neurological disease other than Parkinson's disease (i.e. multiple sclerosis, stroke) that impacts motor or cognitive function
4. Uncontrolled cardiovascular risk factor such as a current cardiac arrhythmia, uncontrolled hypertension, untreated deep vein thrombosis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data is being shared.

REFERENCES:
- [Derived] Koop MM, Rosenfeldt AB, Berki V, Bazyk A, Davidson S, Malan NS, Nagel S, Walter BL, Liao JY, Alberts JL. A novel methodological approach to understanding the cortical and subcortical effects of aerobic exercise in Parkinson's disease. Front Hum Neurosci. 2025 Oct 20;19:1657049. doi: 10.3389/fnhum.2025.1657049. eCollection 2025. PMID 41189627

RESULTS

PARTICIPANT FLOW:
Groups:
- FE Then VE: People with Parkinson's disease (PD) who have undergone DBS surgery and utilize the Percept system completed two stationary bike exercise sessions: forced exercise (FE) and voluntary exercise (VE). FE is a mode of high intensity exercise in which voluntary exercise rate is augmented, but not replaced. VE is standard stationary cycling. The order in which the exercise sessions were completed was randomized. This group of participants was randomized to FE as their first exercise session, and VE as their second exercise session. Participants completed the sessions OFF PD medication. The finger-tapping portion of the MDS-UPDRS III, force-tracking data, and local field potentials (LFPs) were collected before and after exercise sessions. Because all participants completed both exercise interventions, the baseline characteristics and outcome measures are reported by intervention and not by randomization.
- VE Then FE: People with Parkinson's disease (PD) who have undergone DBS surgery and utilize the Percept system completed two stationary bike exercise sessions: forced exercise (FE) and voluntary exercise (VE). FE is a mode of high intensity exercise in which voluntary exercise rate is augmented, but not replaced. VE is standard stationary cycling. The order in which the exercise sessions were completed was randomized. This group of participants was randomized to VE as their first exercise session, and FE as their second exercise session. Participants completed the sessions OFF PD medication. The finger-tapping portion of the MDS-UPDRS III, force-tracking data, and local field potentials (LFPs) were collected before and after exercise sessions. Because all participants completed both exercise interventions, the baseline characteristics and outcome measures are reported by intervention and not by randomization.
Period: First Intervention (1 day)
Arm/Group | FE Then VE | VE Then FE
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout (at least 1 day)
Arm/Group | FE Then VE | VE Then FE
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (1 day)
Arm/Group | FE Then VE | VE Then FE
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Arm: People with Parkinson's disease (PD) who have undergone DBS surgery and utilize the Percept system completed two stationary bike exercise sessions: forced exercise (FE) and voluntary exercise (VE). FE is a mode of high intensity exercise in which voluntary exercise rate is augmented, but not replaced. VE is standard stationary cycling. The order in which the exercise sessions were completed was randomized. Participants completed the sessions OFF PD medication. The finger-tapping portion of the MDS-UPDRS III, force-tracking data, and local field potentials (LFPs) were collected before and after exercise sessions.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Duration of Parkinson's disease [Mean (Standard Deviation); unit: years] | 9.2 (3.8)
Time since DBS placement [Median (Full Range); unit: years] | 1.5 [0.5 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Finger Tapping
Description: Finger tapping portion of the the Movement Disorders Society-Unified Parkinson's Disease Rating Scale subscale III (MDS-UPDRS III). The MDS-UPDRS III assesses motor function in Parkinson's disease using eighteen items scored on a 0-4 scale resulting in a score ranging from 0-72. A higher score (larger number) indicates more motor symptoms. For this outcome, item number 4 (finger tapping rated 0-4) for the participant's dominant hand in the MDS-UPDRS III was analyzed.
Time Frame: Pre- and Post-Exercise
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Experimental Arm
Number analyzed (Participants) | 15
score on a scale
  ON DBS | 3 [2 to 3]
  Pre-FE OFF DBS | 3 [3 to 4]
  Post-FE OFF DBS | 3 [2.5 to 3.5]
  Pre-VE OFF DBS | 3 [3 to 4]
  Post-VE OFF DBS | 3 [2.5 to 3]

2. Primary Outcome: Force Tracking
Description: Participants were required to modulate the precision grip force of their dominant hand to match a target trajectory on a computer screen. Time within range is the percentage of the trial that participants were within 5% of the target force, with higher values indicating improved accuracy.
Time Frame: Pre- and Post-Exercise
Population: Due to a technology error, data is unavailable for the first 2 participants. Complete data is available for 13 participants
Measure: Mean (Standard Deviation); unit: percentage of time within range
Arm/Group | Experimental Arm
Number analyzed (Participants) | 13
percentage of time within range
  ON DBS | 43.3 (23.5)
  Pre-FE OFF DBS | 44.9 (20.4)
  Post-FE OFF DBS | 41.5 (21.4)
  Pre-VE OFF DBS | 43.0 (16.5)
  Post-VE OFF DBS | 41.9 (16.3)

3. Primary Outcome: Local Field Potential
Description: Normalized beta band activity (the change in beta power relative to a resting baseline) is reported as the mean across voluntary exercise (VE) and forced exercise (FE) sessions. The ON DBS condition was not tested for this outcome measure.
Time Frame: Pre- and Post-Exercise
Population: All 15 participants (30 exercise sessions, 1 FE and 1 VE per participant) were included in the analysis, but only 28 of the 30 total exercise sessions were included due to a technology error during 2 of the sessions.
Measure: Mean (Standard Deviation); unit: percent power relative to baseline
Arm/Group | Experimental Arm
Number analyzed (Participants) | 15
percent power relative to baseline
  Pre-FE OFF DBS Left STN | 100.0 (0.0)
  Pre-FE OFF DBS Right STN | 100.0 (0.0)
  Post-FE OFF DBS Left STN | 131.0 (38.3)
  Post-FE OFF DBS Right STN | 120.5 (34.0)
  Pre-VE OFF DBS Left STN | 100.0 (0.0)
  Pre-VE OFF DBS Right STN | 100.0 (0.0)
  Post-VE OFF DBS Left STN | 118.8 (27.2)
  Post-VE OFF DBS Right STN | 110.8 (27.7)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 days.
Groups:
- Pre-FE: Outcome assessed pre-forced exercise. All participants completed a forced exercise (FE) and voluntary exercise (VE) session on a stationary bike. The order of the exercise sessions was randomized for each participant. Outcome measures were assessed Pre- and Post-Exercise. Exercise sessions and outcome measures were performed OFF PD medication.
- Post-FE: Outcome assessed post-forced exercise. All participants completed a forced exercise (FE) and voluntary exercise (VE) session on a stationary bike. The order of the exercise sessions was randomized for each participant. Outcome measures were assessed Pre- and Post-Exercise. Exercise sessions and outcome measures were performed OFF PD medication.
- Pre-VE: Outcome assessed pre-voluntary exercise. All participants completed a forced exercise (FE) and voluntary exercise (VE) session on a stationary bike. The order of the exercise sessions was randomized for each participant. Outcome measures were assessed Pre- and Post-Exercise. Exercise sessions and outcome measures were performed OFF PD medication.
- Post-VE: Outcome assessed post-voluntary exercise. All participants completed a forced exercise (FE) and voluntary exercise (VE) session on a stationary bike. The order of the exercise sessions was randomized for each participant. Outcome measures were assessed Pre- and Post-Exercise. Exercise sessions and outcome measures were performed OFF PD medication.
Arm/Group | Pre-FE | Post-FE | Pre-VE | Post-VE
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT05905302/Prot_SAP_000.pdf